CLINICAL TRIAL: NCT04831996
Title: A Phase 1, Open-Label Study to Evaluate the Pharmacokinetics and Safety of Parsaclisib in Participants With Normal Renal Function and Participants With Renal Impairment
Brief Title: To Evaluate the Safety, and Pharmacokinetics of Parscaclisib in Participants With Normal Renal Function and Renal Impairment.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: INCB 50465-109
Record Dates: First submitted 2021-04-02; First posted 2021-04-05 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2022-08

CONDITIONS: Advanced Malignancies
MeSH Terms: interventions — parsaclisib

STUDY DESIGN:
Masking Description: Open Label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Treat Group 1 : Normal Renal Function (Experimental): eGFR: ≥ 90 mL/min/1.73 m^2
  Interventions: Drug: parsaclisib
- Treat Group 2 : Mild Renal Impairment (Experimental): eGFR: 60-89 mL/min/1.73 m^2
  Interventions: Drug: parsaclisib
- Treat Group 3 : Moderate Renal Impairment (Experimental): eGFR: 30-59 mL/min/1.73 m^2
  Interventions: Drug: parsaclisib
- Treat Group 4 : Severe Renal Impairment (Experimental): eGFR: 15-29 mL/min/1.73 m^2 and not on Hemo Dialysis
  Interventions: Drug: parsaclisib
- Treat Group 5 : Kidney Failure (Experimental): eGFR: < 15 mL/min/1.73 m^2 on Hemo Dialysis
  Interventions: Drug: parsaclisib

INTERVENTIONS:
Drug: parsaclisib — parsaclisib will be administered orally after 8 hours of fasting.
  Other Names: INCB050465

SUMMARY:
The purpose of the study is to evaluate the pharmacokinetics and safety of parsaclisib in participants With normal renal function and participants with renal impairment.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be classified at screening by renal function based on eGFR as calculated by the MDRD formula and requirement for HD (Group 5).
* Participants eligible for Group 5 with ESRD have received HD for at least 3 months prior to screening.
* Participants eligible for Group 1 should be in good health as determined by no clinically significant deviations from normal for medical history, physical examination, vital signs, 12-lead ECGs, or clinical laboratory determinations at screening or Day -1.
* Participants eligible for Groups 2 through 5 may have medical findings consistent with their degree of renal dysfunction.
* Participants with abnormal findings considered not clinically significant by the medical monitor or investigator are eligible.

  0Body mass index within the range 18.0 to 40.0 kg/m2 (inclusive) at screening.
* Willingness to avoid pregnancy or fathering children.
* Ability to swallow and retain oral medication.

Exclusion Criteria:

* History of uncontrolled or unstable cardiovascular, respiratory, hepatic, gastrointestinal, endocrine, hematopoietic, psychiatric, and/or neurological disease within 6 months of screening. Evidence of rapidly deteriorating renal function.
* Participants who have a current, functioning organ transplant or have a scheduled organ transplant within 6 weeks after check-in.
* History of malignancy within 5 years of screening, with the exception of cured basal cell carcinoma, squamous cell carcinoma of the skin, ductal carcinoma in situ, or Gleason 6 prostate cancer.
* History of clinically significant gastrointestinal disease or surgery (cholecystectomy and appendectomy are allowed) that could impact the absorption of study drug.
* Participants eligible for Group 1 who have a history of renal disease or renal injury as indicated by an abnormal, clinically significant renal function profile at screening or Day -1.
* Participants eligible for Groups 2 through 5 who have had a change in disease status within 30 days of screening, as documented by the participant's medical history, deemed clinically significant by the investigator.
* History or current diagnosis of uncontrolled or significant cardiac disease indicating significant risk of safety for participation in the study.
* Any major surgery within 4 weeks of screening.
* Donation of blood to a blood bank within 4 weeks of screening (within 2 weeks for plasma only).
* Blood transfusion within 4 weeks of Day -1 (for Groups 1 through 4) or Period 1, Day
* 1 (Group 5).
* Chronic or current active infectious disease requiring systemic antibiotic, antifungal, or antiviral treatment.
* Positive test for HBV (HBsAg, HBsAg antibody, and hepatitis B core antibody), HCV (HCV antibody), or HIV. Participants whose results are compatible with prior immunization for HBV may be included at the discretion of the investigator.

Participants eligible for Group 1 who have used tobacco- or nicotine-containing products within 6 months of screening.

* Participants eligible for Groups 2 through 5 who smoke > 10 cigarettes per day or equivalent use of other tobacco- or nicotine-containing products and are unwilling to refrain from tobacco or nicotine use on dosing days and abide by CRU restrictions.
* Positive breath test for ethanol or positive urine or serum screen for drugs of abuse that is not otherwise explained by permitted concomitant medications.
* Current treatment or treatment within 30 days or 5 half-lives (whichever is longer) of study drug administration with another investigational medication or current enrollment in another investigational drug study.
* Current treatment or treatment within 30 days or 5 half-lives (whichever is longer) of study drug administration with strong or moderate inducer or inhibitor of CYP3A4, P-gp,or BCRP.
* For participants eligible for Group 1, use of prescription drugs within 14 days of study drug administration or nonprescription medications/products (including vitamins, minerals, and phytotherapeutic/herbal/plant-derived preparations) within 7 days of study drug administration. However, occasional paracetamol, ibuprofen, and standard-dose vitamins are permitted.
* For participants eligible for Groups 2 through 5, use of prescription drugs within 14 days of study drug administration, with the exception of established therapy for renal disease and the treatment of associated disorders that have been stable for at least 7 days prior to study drug administration, as approved by the investigator and in consultation with the sponsor's medical monitor.
* Current or recent history (within 30 days before screening) of a clinically significant bacterial, fungal, parasitic, or mycobacterial infection, or currently receiving systemic antibiotics. Current clinically significant viral infection at screening or check-in.
* History of any significant drug allergy (such as anaphylaxis or hepatotoxicity) deemed clinically relevant by the investigator.
* Inability to undergo venipuncture or tolerate venous access.
* Participants eligible for Group 5 that are not expected to continue HD treatment for the duration of the study.
* Receipt of live (including attenuated) vaccines or anticipation of need for such a vaccine during the study (Note: nonlive or inactivated vaccines are allowed up to 2 weeks prior to the first dose of study drug).
* Known hypersensitivity or severe reaction to parsaclisib or excipients of parsaclisib.
* History of alcoholism within 3 months of screening.
* Women who are pregnant or breastfeeding.

Ages: 18 Years to 82 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2021-05-04 (Actual); Primary Completion 2022-07-08 (Actual); Study Completion 2022-07-08 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics Parameter Groups1-4 : Cmax of parsaclisib | 4 Days
  Maximum Observed Plasma Concentration of parsaclisib
Pharmacokinetics Parameter Groups 1-4 : AUC 0-∞ of parsaclisib | 4 Days
  Area Under the Concentration-time Curve From 0 to Infinity of parsaclisib
Pharmacokinetics Parameter Groups 1-4 : AUC(0-t) of parsaclisib | 4 Days
  Area Under the concentration- time curve up to the last measurable concentration of parsaclisib
Pharmacokinetics Parameter Group 5: Cmax of parsaclisib | 4 Days for period 1 and 2
  Maximum Observed Plasma Concentration of parsaclisib
Pharmacokinetics Parameter Group 5 : AUC 0-∞ of parsaclisib | 4 Days for period 1 and 2
  Area Under the Concentration-time Curve From 0 to Infinity of parsaclisib
Pharmacokinetics Parameter Group 5: AUC(0-t) of parsaclisib | 4 Days for period 1 and 2
  Area Under the concentration- time curve up to the last measurable concentration of parsaclisib

SECONDARY OUTCOMES:
Number of Treatment Emergent Adverse Events (TEAE) Groups 1-4 | up to 11 Days
  Adverse events reported for the first time or worsening of a pre-existing event after first dose of study drug/treatment.
Pharmacokinetics Parameter Groups 1-4 : tmax of parsaclisib | 4 Days
  Time to reach maximum plasma concentration of parsaclisib
Pharmacokinetics Parameter Groups 1-4 : t1/2 of parsaclisib | 4 Days
  Apparent terminal phase disposition half-life of parsaclisib
Pharmacokinetics Parameter Groups 1-4 : CL/F of parsaclisib | 4 Days
  Oral dose clearance of parsaclisib
Pharmacokinetics Parameter Groups 1-4 : Vz/F of parsaclisib | 4 Days
  Apparent oral dose volume of distribution of parsaclisib
Pharmacokinetics Parameter Group 5 : tmax of parsaclisib | 4 Days for period 1 and 2
  Time to reach maximum plasma concentration of parsaclisib
Pharmacokinetics Parameter Group 5 : t1/2 of parsaclisib | 4 Days for period 1 and 2
  Apparent terminal phase disposition half-life of parsaclisib
Pharmacokinetics Parameter Group 5 : CL/F of parsaclisib | 4 Days for period 1 and 2
  Oral dose clearance of parsaclisib
Pharmacokinetics Parameter Group 5 : Vz/F of parsaclisib | 4 Days for period 1 and 2
  Apparent oral dose volume of distribution of parsaclisib
Pharmacokinetics Parameter Group 5 during Dialysis - : AUC1-5 of parsaclisib | 4 Days for period 1 and 2
  Area Under the Concentration-time Curve From 1 to 5 hrs. of parsaclisib
Number of Treatment Emergent Adverse Events (TEAE) Group 5 | up to 18 Days
  Adverse events reported for the first time or worsening of a pre-existing event after first dose of study drug/treatment.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Orange County Research Center, Tustin, California
  - Clinical Pharmacology of Miami, Hialeah, Florida
  - Orlando Clinical Research Center, Orlando, Florida
  - Prism Research, Saint Paul, Minnesota

IPD SHARING:
Plan to Share IPD: Yes
Incyte shares data with qualified external researchers after a research proposal is submitted. These requests are reviewed and approved by a review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  The trial data availability is according to the criteria and process described on https://www.incyte.com/our-company/compliance-and-transparency
Supporting Information: Study Protocol
Time Frame: Data will be shared after the primary publication or 2 years after the study has ended for market authorized products and indications.
Access Criteria: Data from eligible studies will be shared with qualified researchers according to the criteria and process described in the Data Sharing section of the www.incyteclinicaltrials.com website. For approved requests, the researchers will be granted access to anonymized data under the terms of a data sharing agreement.
URL: https://www.incyte.com/our-company/compliance-and-transparency